CLINICAL TRIAL: NCT01381458
Title: Differences in the Risk of Re-hospitalization and Other COPD-related (Chronic Obstructive Pulmonary Disease) Exacerbations and Costs for Patients Receiving Fluticasone Propionate-salmeterol Xinafoate Combination 250/50mcg (FSC) Versus Anticholinergics [i.e. Tiotropium (TIO) and Ipratropium or Combination Ipratropium-albuterol (IPR) Post-hospitalization or ED Visit for the Treatment of COPD.
Brief Title: Risk of Re-Hospitalization in Patients With Chronic Obstructive Pulmonary Disease (COPD) Post Exacerbation
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113899
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD patients receiving pharmacotherapy: COPD patients age 40 years and older receiving pharmacotherapy to treat their COPD and an index event of COPD hospitalization or ER visit.
  Interventions: Drug: FSC; Drug: ACs

INTERVENTIONS:
Drug: FSC — fluticasone propionate / salmeterol xinofoate combination
  Other Names: Advair (tm)
Drug: ACs — tiotropium alone, ipratropium alone, or in combination with albuterol

SUMMARY:
This retrospective database study will assess differences in the risk of re-hospitalization and other COPD-related exacerbations and costs for patients receiving fluticasone propionate/salmeterol xinafoate combination 250/50 (FSC) versus anticholinergics [i.e. tiotropium (TIO) and ipratropium or combination ipratropium-albuterol (collectively referred to as ipratropium - IPR)] post-hospitalization or Emergency Department (ED) visit for the treatment of COPD.

This is a hypotheses testing study. Associations are compared between FSC and AC cohorts.

Hypotheses for the primary outcome and key secondary outcomes are presented below:

Specifically the study hypotheses for the primary outcome being tested were:

Ho: There is no difference in risk of COPD-related hospitalization between FSC and AC Ha: There is a difference in risk of COPD-related hospitalization between FSC and AC

Hypothesis for the key secondary outcome of COPD-related costs that was tested was:

Ho: There is no difference in COPD-related costs between FSC and AC Ha: There is a difference in COPD-related costs between FSC and AC

DETAILED DESCRIPTION:
Managed care patients (aged >40 years) who were fluticasone propionate/salmeterol xinafoate combination (FSC)-naive in the 12 months pre-index period. The index-date was the date of discharge of the index Chronic Obstructive Pulmonary Disease (COPD)-related hospitalization/Emergency Department (ED) visit. Eligible patients were required to newly initiate or switch to drug therapy with FSC or ipratropium (IPR) / tiotropium (TIO) during the identification period (01/01/2004 to 01/31/2008) to treat COPD. Patients who switched to another maintenance medication or had an exacerbation in the treatment assessment period (30-days post-index date) were excluded from the study. Follow-up period was 12 months post treatment assessment period. Patients classified as being on FSC 250/50 versus anticholinergics (TIO, IP or IPR). Examined risk of COPD-related exacerbations such as hospitalizations, emergency department (ED) visits, COPD-related physician/outpatient visit with oral corticosteroid (OCS) or antibiotic prescription (ABX) within 5 days of physician/outpatient visit and COPD-related medical, pharmacy, and total healthcare costs in follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* ≥40 years of age at index discharge date
* Continuous health plan eligibility in the pre-index, treatment assessment, and follow-up periods
* Absence of other fluticasone propionate -salmeterol xinafoate doses or combination product of budesonide-formoterol anytime during pre-index, treatment assessment, and follow-up periods

Exclusion Criteria:

* COPD-related exacerbation during the treatment assessment period
* Any therapy change, which was defined as switching or augmenting index therapy during treatment assessment period
* Absence of comorbid conditions (respiratory cancer, cystic fibrosis, fibrosis due to tuberculosis, bronchiectasis, pneumonociosis, pulmonary fibrosis, pulmonary tuberculosis, and sarcoidosis) during the pre-index, treatment assessment, and follow-up periods

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Managed care patients (aged >40 years) who were FSC naive in the 12 months pre-index period. The index-date was the date of discharge of the index COPD-related hospitalization/ED visit. Eligible patients were required to newly initiate or switch to drug therapy with FSC or IPR/TIO during the identification period (01/01/2004 to 01/31/2008) to treat COPD. Patients who switched to another maintenance medication or had an exacerbation in the treatment assessment period (30-days post-index date) were excluded from the study. Follow-up period was 12 months post treatment assessment period.
Sampling Method: Non-Probability Sample
Enrollment: 1936 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Risk of Hospitalization in COPD patients | January 1, 2003 through March 31, 2009 (up to 6 years)
  Risk of hospitalization was assessed as any hospitalization that was catpured in the follow up period. We required this event to have a primary discharge dx of COPD (ICD-9 code 491.xx, 492.xx, 496.xx) thus assuring it to be COPD-related. a logistic regression model was run to examine this outcome.

SECONDARY OUTCOMES:
Number of COPD exacerbations | January 1, 2003 through March 31, 2009 (up to 6 years)
  Exacerbation rates were assessed between the FSC and AC groups. We examined COPD-related (primary dx of COPD (ICD-9 code 491.xx, 492.xx, 496.xx)) emergency department visits, outpatient visits, outpatient visits accompanied by prescription of oral steroids and antibiotics. A negative binomial regression model was run to examine this outcome.
COPD-related Costs | January 1, 2003 through March 31, 2009 (up to 6 years)
  Mean COPD-related medical costs-, pharmacy costs - and total costs (the sum of medical and pharmacy costs) were calculated. Medical costs included healthcare facility and professional services charges for hospital admissions, ED visits, physician and other outpatient visits, and laboratory, radiology and other outpatient procedures with a primary diagnosis of COPD. Costs were adjusted to 2009 US dollars using the medical care component of the Consumer Price Index (CPI ). A Generalized Linear Model (GLM) with a log-link function was used to assess differences in costs.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline